CLINICAL TRIAL: NCT00882310
Title: A Phase II Study of Gemzar, Taxotere, and Xeloda (GTX) for Adjuvant Pancreatic Cancer
Brief Title: A Study of Gemzar, Taxotere, and Xeloda for Adjuvant Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB4460
Record Dates: First submitted 2009-03-23; First posted 2009-04-16 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Gemzar; Taxotere; Xeloda; GTX
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Docetaxel, Capecitabine GTX (Experimental): GTX - A two week regimen of Gemcitabine at 600 mg/m2 on days 4 and 1, infused over 60 minutes, Docetaxel at 30 mg/m2 on days 4 and 11, infused over 60 minutes and Capecitabine at 1000 mg/m2 (capped at 1000 mg BID days 1-14) followed by one week off for a total of a 21 day cycle. This is repeated for a total of 6 months.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Gemcitabine — Days 4 and 11: gemcitabine 600 mg/m2 over 60 mins intravenous (IV) followed by docetaxel 30 mg/m2 over 60 mins IV
  Other Names: Gemzar
Drug: Docetaxel — Days 4 and 11: gemcitabine 600 mg/m2 over 60 mins intravenous (IV) followed by docetaxel 30 mg/m2 over 60 mins IV
  Other Names: Taxotere
Drug: Capecitabine — Day 1-14: capecitabine at 1000 mg/m2/day divided into 2 doses given two times a day (BID) by mouth (PO) Maximum dose 2000mg/day divided into BID dosing
  Other Names: Xeloda

SUMMARY:
The main purpose of this study will be to evaluate the toxicities as well as the efficacy of a chemotherapy regimen involving the combination of Gemzar, Taxotere, and Xeloda (GTX) in patients with pancreatic cancer, who have undergone complete surgical resection of their tumor. During the screening evaluation, subjects will have a physical exam and medical history taken by either the PI or a Co investigator. In addition, routine blood tests and radiological exams will be performed, to determine eligibility. Following enrollment, patients will receive 8 cycles (1 cycle = 21 days) of GTX treatment over 6 months. During each cycle patients will receive Gemzar and Taxotere on days 4 and 11, through an IV, over the course of approximately 2 hours, and Xeloda will be taken orally for the first 14 days of every cycle. Patients will receive no treatment on days 15 thru 21 of each cycle. During each cycle of treatment patients will have a physical examination, as well as routine blood work. The first scan will be done prior to initiation of treatment, and the next will be done at completion of chemotherapy. A short quality of life questionnaire will also be administered prior to cycle 1 treatment, at the 3-month point, and at the completion of chemotherapy.

DETAILED DESCRIPTION:
The adjuvant treatment of resected pancreatic cancer is currently in flux. Many in the United States continue to use 5FU-based chemotherapy with radiation to the pancreatic bed. Some in the States, and most investigators in Europe, use a 5FU based chemotherapy-alone approach, based on the ESPAC-1 data. Many investigators believe that since gemcitabine is a more active drug in the metastatic setting, it should be moved "up front" in the adjuvant treatment of pancreatic cancer patients. At Columbia, we offer gemcitabine-based treatments with discussions with patients regarding risks, benefits, and limitations in current knowledge. We have usually offered radiation to those with positive margins, and chemotherapy alone to those without. Based on the early studies using gemcitabine, we believe that this will ultimately prove to be a more effective adjuvant drug than 5FU. Some patients have asked for GTX in the adjuvant setting as well, prompting the creation of this trial. Because of concerns about increased toxicity of this regimen, determination of patient safety will be the primary objective of this study, through careful monitoring of adverse events. This trial will be a chemotherapy-only study, offered to those with clean margins of resection.

Taxotere administered "weekly" has activity in a variety of tumor types including breast, lung, ovarian and prostate cancer. Patients with advanced breast cancer, including some who had previously been treated with paclitaxel or anthracyclines, have responded to the weekly administration of Taxotere. The recommended dose of weekly Taxotere is 30-40 mg/m2/week for 6 out of 8 weeks. The same dose intensity can be achieved on a 3 out of 4 week basis. However, this protocol will give drugs 2 out of every 3 weeks, thus dose intensity is less.

Weekly administration of Taxotere is well tolerated and produces substantially less myelosuppression than is observed with standard Taxotere administration every 3 weeks. Acute toxicities are uncommon, as is peripheral neuropathy. Prolonged treatment with weekly Taxotere, may result in chronic toxicities (including, asthenia (fatigue), anemia, edema, excessive lacrimation (epiphora), and onycholysis). Chronic toxicities are most prominent when Taxotere is administered on a continuous weekly basis, i.e., without a break, and are delayed in onset by providing breaks in treatment (for example, treating 6 out of 8 weeks or 3 out of 4 weeks); these chronic toxicities occur at a lower cumulative dose when a continuous weekly schedule of Taxotere is utilized.

Premedication with dexamethasone is recommended for all patients receiving weekly Taxotere therapy to reduce the incidence and severity of fluid retention as well as the severity of hypersensitivity reactions. A variety of dexamethasone schedules have been used in studies with weekly Taxotere. Dexamethasone 4 to 8 mg x 3 doses taken orally the night before, the morning of, and the evening after Taxotere administration appears to be an effective schedule. We have found that a single low dose of 10 mg IV before the Taxotere usually prevents anaphylaxis and the pedal edema associated with this drug.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of pancreas that has been completely resected. Patients may be node negative or node-positive, but must have clean margins of resection.
* Ineligible for other high priority national or institutional studies.
* Time from surgical recovery greater than three weeks, but less than six weeks.
* All radiological evaluations (which must include either CT scans of the chest/abdomen/pelvis or a CT of the chest and a MRI of the abdomen/pelvis) must be performed within 4 weeks prior to the start of study therapy.
* Informed Consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.
* Non pregnant females who are not breast feeding with a negative serum β-HCG test within 1 week of starting the study. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for 6 months after completion of treatment. They must understand the risks of infertility possibly associated with adjuvant treatment.
* Clinical Parameters:

  * Age ≥ 18 to ≤ 75 years old
  * Performance status 0-2 (ECOG)
  * Peripheral Neuropathy must be < grade 1
  * Able to tolerate oral medications
  * Absolute Neutrophil Count > 1,500 ul
  * White Blood Count > 3,000/ul
  * Platelet count > 100,000/ul
  * BUN < 1.5 x ULN
  * Creatinine < 1.5 x ULN
  * Hemoglobin > 8.0 g/dl
  * Serum Albumin > 2.5 mg/dl
  * Total Bilirubin < 3.0 mg/dl
  * AST ≤4.0 x ULN
  * ALT ≤4.0 x ULN
  * Alkaline Phosphatase ≤4.0 x ULN]
  * CA 19-9 should be normal post surgery. Can still be put on protocol with elevation if clinically significant for inflammation or infection, not cancer

Exclusion Criteria:

* Prior chemotherapy for their pancreatic cancer or radiation to the area of the tumor.
* Prior malignancies in last 5 years other than curatively treated carcinoma in-situ of any site in the body.
* Serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g., serious infection).
* Patients with compromised immune systems are at increased risk of toxicity and lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients are excluded from the study.
* Any prior investigational agent/therapy or any investigational agent/therapy while on protocol.
* Hypersensitivity: Patients with a history of severe hypersensitivity reaction to Taxotere® or other drug formulated with polysorbate 80 will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Oberstein, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Docetaxel, Capecitabine GTX
Started | 37
Completed | 15
Not Completed | 22
Not completed — Screen Failure | 10
Not completed — Never received treatment | 1
Not completed — Death | 6
Not completed — Progression of disease | 4
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Docetaxel, Capecitabine GTX
Number analyzed (Participants) | 37
Age, Customized [Number; unit: participants]
  40-49 | 5
  50-59 | 8
  60-69 | 17
  70-79 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 4
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experience Dose Limiting Toxicities (DLTs)
Description: Safety of the GTX regimen in patients with resected pancreatic cancer, using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
  Data was not analyzed because original PI left institution before data analysis was completed.
Time Frame: At days 4, 11, and follow-up.
Arm/Group | Gemcitabine, Docetaxel, Capecitabine GTX
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Death
Description: Median recurrence free survival in patients with non-metastatic, resected pancreatic cancer treated with adjuvant GTX.
  Data was not analyzed because original PI left institution before data analysis was completed.
Time Frame: At 6 months (following completion of treatment), and then every 3 months for the first 2 years. After the first 2 year, annually.
Arm/Group | Gemcitabine, Docetaxel, Capecitabine GTX
Number analyzed (Participants) | 0

3. Secondary Outcome: Score on FACT-Hep (Version 4)
Description: Quality of life score of patients treated with the adjuvant GTX regimen using, the FACT-Hep (Version 4), a sensitive measure of quality of life.
  Data was not analyzed because original PI left institution before data analysis was completed.
Time Frame: Prior to starting treatment, after 3 months of treatment, and at the end of study visit.
Arm/Group | Gemcitabine, Docetaxel, Capecitabine GTX
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: AE data was collected on 26 subjects (out of 37 subjects, 10 were screen failures and 1 was not treated).
Groups:
- Gemcitabine, Docetaxel, Capecitabine GTX: GTX - A two week regimen of Gemcitabine at 600 mg/m2 on days 4 and 1, infused over 60 minutes, Docetaxel at 30 mg/m2 on days 4 and 11, infused over 60 minutes and Capecitabine at 1000 mg/m2 (capped at 1000 mg BID days 1-14) followed by one week off for a total of a 21 day cycle. This is repeated for a total of 6 months.
  AE data was collected on 26 subjects (out of 37 subjects, 10 were screen failures and 1 was not treated).
Arm/Group | Gemcitabine, Docetaxel, Capecitabine GTX
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Docetaxel, Capecitabine GTX (N=26)
Progression of Disease leading to death (General disorders) | 5 (5)
Death of unknown reason (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Docetaxel, Capecitabine GTX (N=26)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes